CLINICAL TRIAL: NCT00786487
Title: Training Effects on Skeletal Muscle Fatty Acid Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 0804M29862; pending (Other Grant/Funding Number: pending)
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Healthy Volunteers
Keywords: insulin resistance; lipid metabolism; lipid infusion; glycerol infusion; skeletal muscle; diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus | interventions — soybean oil, phospholipid emulsion; Glycerol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- lipid trained (Experimental): 20% lipid infusion in trained subjects
  Interventions: Drug: 20% lipid infusion
- glycerol trained (Active Comparator): glycerol infusion into trained subjects
  Interventions: Drug: glycerol
- lipid untrained (Experimental): lipid infusion into untrained subjects
  Interventions: Drug: 20% lipid infusion
- glycerol untrained (Active Comparator): glycerol infusion into untrained subjects
  Interventions: Drug: glycerol

INTERVENTIONS:
Drug: 20% lipid infusion — 1.5 ml/min for 6 hours
  Other Names: Intralipid; triglyceride infusion; lipid infusion; fat infusion
  Arms: lipid trained; lipid untrained
Drug: glycerol — glycerol infusion (2.25 g/100ml) will be administered at 1.5 ml/min,
  Other Names: Control infusion; glycerol infusion
  Arms: glycerol trained; glycerol untrained

SUMMARY:
We are interested in how skeletal muscle processes fat and how this may affect insulin resistance. This is an important question since insulin resistance predates and predicts type 2 diabetes. We know that if pharmaceutical grade fat is infused into people, they develop insulin resistance. Likewise, we would like to infuse pharmaceutical grade fat into trained subjects, believing that trained subjects will have less insulin resistance, less decline in muscle energy function, and less accumulation of fat metabolites than untrained subjects. For comparing the effects of the pharmaceutical grade fat infusion, we will also have a group of trained and untrained subjects given a control (glycerol) infusion. Glycerol is basically the same as pharmaceutical grade fat infusion without the fat component.

DETAILED DESCRIPTION:
We are interested in how skeletal muscle processes fat and its effect on insulin resistance. This is an important question since insulin resistance predates and predicts type 2 diabetes. We know that if pharmaceutical grade lipid is infused into people, they develop insulin resistance. Thus, we would like to infuse pharmaceutical grade lipid into trained subjects, believing that trained subjects will develop less insulin resistance, less decline in muscle energy function, and less accumulation of fat metabolites than untrained subjects. For comparing the effects of the pharmaceutical grade fat infusion, we will also have a group of trained and untrained subjects given a control (glycerol) infusion. Glycerol is basically the same as pharmaceutical grade lipid infusion without the lipid component.

Three visits will be required. The first visit will involve measurement of fitness. A second visit will involve measurement of insulin resistance. The third visit will involve an inpatient stay, with a six hour infusion either the lipid or glycerol. Three muscle biopsies (before, during and after) will be take in conjunction with the infusion.

ELIGIBILITY:
Inclusion Criteria:

* Regardless of training status, age range will be from age 18 to 45. We will be limiting the upper age range because increased age is associated with sarcopenia and alteration of fiber type 29 and we would like to limit the confounding effects of age.
* We will define the lean group by a BMI of < 25 kg/m2. Weight must be stable [+/- 5 pounds] for at least the three months prior to the study for all participants.
* The untrained subjects must not be engaged in a regular exercise program (< 30 minutes regular exercise over 1 week).
* The trained subjects should be participating in regular running exercise (> 45 min/day, ≥ 5 days/week) and preferably be currently or recently participating in competitions (within 2 years).

Exclusion Criteria:

* Regardless of training status, subjects must not be on medications that may affect lipid levels, specifically lipid lowering agents, birth control pills or diuretics.
* The subjects should not be on a high fat diet (> 45% fat) as measured by a screening questionnaire. We will also administer a PAR-Q questionnaire (attached) to establish whether the subject will be safe for exercise testing. - The female subjects must not be pregnant. A pregnancy test will be performed prior to all study visits.
* If screening TG are > 300 (based on 1st visit results) or fasting glucose > 100 (based on 1st visit results), the subjects will be excluded.
* If the subject is allergic to eggs (used in lipid emulsions), soybeans(used in lipid emulsions), or lipid emulsions the subject will be excluded from the study.
* Subjects taking anti-platelet agents (if anti-platelet agent cannot be held for seven days) and subjects taking anticoagulation therapy will be excluded.
* Subjects with clinically significant medical issues or a history of hematologic (platelets < 100), hepatic (LFTs > 2X nl), renal (Cr > 1.5), pulmonary, or cardiac abnormalities (including abnormal EKG) will also be excluded.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2009-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa S Chow, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Chow LS, Seaquist ER, Eberly LE, Mashek MT, Schimke JM, Nair KS, Mashek DG. Acute free fatty acid elevation eliminates endurance training effect on insulin sensitivity. J Clin Endocrinol Metab. 2012 Aug;97(8):2890-7. doi: 10.1210/jc.2012-1515. Epub 2012 May 25. PMID 22639293

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: we had anticipated enrollment of 36 subjects but ended up finishing the study with 33 subjects
Period: Overall Study
Arm/Group | Lipid Trained | Glycerol Trained | Lipid Untrained | Glycerol Untrained
Started | 10 | 7 | 9 | 7
Completed | 10 | 7 | 9 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lipid Trained | Glycerol Trained | Lipid Untrained | Glycerol Untrained | Total
Number analyzed (Participants) | 10 | 7 | 9 | 7 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 7 | 9 | 7 | 33
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (6) | 24 (3) | 21 (2) | 21 (2) | 23 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 4 | 3 | 15
  Male | 5 | 4 | 5 | 4 | 18
Region of Enrollment [Number; unit: participants]
  United States | 10 | 7 | 9 | 7 | 33
insulin sensitivity [Mean (Standard Deviation); unit: M value] | 13.5 (3.5) | 12 (3) | 7 (1.6) | 9 (3) | 10.7 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity as Measured by Hyperinsulinemic Euglycemic Clamp at a Single Time Point (6 Hrs) After Intralipid or Glycerol Infusion
Description: Insulin sensitivity (M value: Glucose infusion rate/kg FFM/min)measured at single time point 6 hours after initiating either intralipid or glycerol infusion)
Time Frame: at 6 hours after starting lipid/glycerol infusion
Measure: Mean (Standard Deviation); unit: M value
Arm/Group | Lipid Trained | Glycerol Trained | Lipid Untrained | Glycerol Untrained
Number analyzed (Participants) | 10 | 7 | 9 | 6
M value | 8 (3) | 12 (2) | 6 (2) | 11 (4)
Statistical Analysis 1: Comparison: Lipid Trained vs Glycerol Trained; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Lipid Untrained vs Glycerol Untrained; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Lipid Trained | Glycerol Trained | Lipid Untrained | Glycerol Untrained
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7 | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 1/10 | 1/7 | 0/9 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lipid Trained (N=10) | Glycerol Trained (N=7) | Lipid Untrained (N=9) | Glycerol Untrained (N=6)
numbness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — slight skin numbness at site of muscle biopsy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No